CLINICAL TRIAL: NCT01485692
Title: Safety and Efficacy of Four Intramuscular Interventions for the Management of Acute Psychomotor Agitation
Brief Title: Four Interventions in the Management of Psychomotor Agitation, Safety and Efficacy Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Celia Mantovani, Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UE0001
Record Dates: First submitted 2011-11-28; First posted 2011-12-05 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2009-02

CONDITIONS: Psychomotor Agitation
Keywords: Violence; Aggression; Psychiatric emergencies; Psychomotor agitation; Violent patient
MeSH Terms: conditions — Psychomotor Agitation; Aggression | interventions — Haloperidol; Midazolam; Olanzapine; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ziprasidone injection (Active Comparator): ziprasidone injection after baseline measures of agitation, could be repeated twice, if necessary, between the 90 minutes of the observation
  Interventions: Drug: Ziprasidone
- haloperidol + midazolam, injection (Active Comparator): Haloperidol plus midazolam injection, after baseline measures of agitation,allowed to be repeated twice over the 90 minutes period of observation
  Interventions: Drug: haloperidol + midazolam
- haloperidol + promethazine, injection (Active Comparator): haloperidol + promethazine injection after baseline measures of agitation, could be repeated after 30 minutes, and once more, if necessary, in the 90 minutes period of observation
  Interventions: Drug: haloperidol+promethazine
- olanzapine, injection (Active Comparator): olanzapine, 10mg, intramuscular injection after baseline measures of agitation, could be repeated twice if necessary, between the 90 minutes of observation
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: haloperidol+promethazine — haloperidol, 2,5mg plus promethazine,25mg, intramuscular injection after baseline measures of agitation, could be repeated twice, if necessary, in the 90 minutes period of observation
  Arms: haloperidol + promethazine, injection
Drug: haloperidol + midazolam — haloperidol, 2,5mg plus midazolam, 7,5 mg, intramuscular injection after baseline measures of agitation, could be repeated twice, if necessary, between the 90 minutes period of observation
  Arms: haloperidol + midazolam, injection
Drug: olanzapine — olanzapine, 10mg, intramuscular injection, after baseline measures of agitation, could be repeated twice, if necessary, between the 90 minutes of observation
  Arms: olanzapine, injection
Drug: Ziprasidone — ziprasidone, 10 mg, intramuscular injection after baseline measures of agitation, could be repeated twice, if necessary, between the 90 minutes period of observation
  Arms: ziprasidone injection

SUMMARY:
This study aims to evaluate the efficacy and safety of four options of medications in the management of acute psychomotor agitation,or violence and aggression situations in health services. All of the treatment options are already approved and currently used for this purpose. The options are: haloperidol plus midazolam, haloperidol plus promethazine, olanzapine and ziprasidone. The investigators hypothesized that all treatment options are effective in the treatment of acute agitation, but the combination haloperidol plus promethazine could elicit more adverse affects than the others.

ELIGIBILITY:
Inclusion Criteria:

* patients featuring psychomotor agitation, with clinical need for intramuscular injection

Exclusion Criteria:

* delirium, severe or unstable general medical condition, previous history of severe adverse effects with one of the treatment options

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction in the agitation score | 90 minutes
  Agitation scores were evaluated through two previously validated specific scales: ACES ( Agitation Calmness Evaluating Scale) and PANSS-EC ( Positive and Negative Symptoms Scale- Excited Component). The measure was collected by a blind rater at baseline and the subsequent measures aimed to evaluate the drug effect over agitation scores.

SECONDARY OUTCOMES:
Adverse effects | 12,24 hours after baseline
  Aiming to evaluate the occurrence of adverse effects in the 24 hours period of observation after administrating the first injection (Baseline), an exert from the UKU scale (Ugvalg klinisk Undersgelser Side Effect Scale )was applied by a blind rater, to evaluate the presence and intensity of possible side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Celia Mantovani, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina de Ribeirão Preto, USP, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Mantovani C, Labate CM, Sponholz A Jr, de Azevedo Marques JM, Guapo VG, de Simone Brito dos Santos ME, Pazin-Filho A, Del-Ben CM. Are low doses of antipsychotics effective in the management of psychomotor agitation? A randomized, rated-blind trial of 4 intramuscular interventions. J Clin Psychopharmacol. 2013 Jun;33(3):306-12. doi: 10.1097/JCP.0b013e3182900fd6. PMID 23609398